CLINICAL TRIAL: NCT02706470
Title: A Randomized, Controlled Trial of Cyclosporin A for Women With Unexplained Recurrent Miscarriage
Brief Title: Use of Cyclosporin A for the Treatment of Recurrent Miscarriage
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiangfeng Ye, MD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013SY034
Record Dates: First submitted 2016-02-02; First posted 2016-03-11 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Miscarriage, Recurrent
Keywords: recurrent miscarriage; immunology
MeSH Terms: conditions — Abortion, Habitual | interventions — Cyclosporine; Dydrogesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporin A (Experimental): Patients allocated to Cyclosporin A group will receive oral Cyclosporin A in a dose of 50 mg three times a day for 20-30 days in early pregnancy.
  Interventions: Drug: Cyclosporin A
- Dydrogesterone (Active Comparator): Patients allocated to dydrogesterone group will receive oral dydrogesterone in a dose of 10 mg three times a day for 30 days in early pregnancy.
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Cyclosporin A — Patients will receive oral CsA in a dose of 50mg three times a day for 20-30 days since the occurrence of positive result in human chorionic gonadotropin (HCG) test in urine and 14 consecutive days of elevated basal body temperature. The dosage of CsA will be adjusted according to baseline and peak value of CsA blood concentration. If the baseline blood concentration of CsA is lower than 40ng/ml or the peak blood concentration of CsA is lower than 500ng/ml, the dosage of CsA will be increased to 75 mg three times a day.
  Arms: Cyclosporin A
Drug: Dydrogesterone — Patients will receive oral dydrogesterone 10 mg three times a day for 30 days since the occurrence of positive result in HCG test in urine and 14 consecutive days of elevated basal body temperature.
  Other Names: Duphaston
  Arms: Dydrogesterone

SUMMARY:
The purpose of this study is to determine whether Cyclosporin A (CsA) - an immunosuppressant drug - in early pregnancy will reduce the risk of miscarriage in women who had a history of unexplained recurrent miscarriages, as compared with that treated with Dydrogesterone-an active comparator. The hypothesis is based on the evidence found in vitro and in vivo experiments that CsA can induce maternal-fetal tolerance so that it may reduce the risk of miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Both the woman and her husband agree to participate and sign the informed consent form.
* Have a history of two or more unexplained recurrent miscarriages.
* Spontaneous conception.
* Gestational age less than 5 weeks.
* Have a normal menstrual cycle (>=23 and <=35 days) and biphasic pattern of basal body temperature before pregnancy.
* No significant chromosomal aberrations in the couple.
* Semen quality tests show not apparent abnormalities in husband

Exclusion Criteria:

* Age below 18 or above 41 years at conception.
* Present pregnancy is a result of donor insemination or egg donation.
* Significant uterine anomalies detected by ultrasonography, hysterosalpingography, or hysteroscopy.
* Contraindications of CsA (e.g. severe infectious diseases, tumor or immunodeficiency) or Dydrogesterone.
* Smoking more than 20 daily.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Up to 36 months
  The difference in the live birth rates between patients with recurrent miscarriage assigned oral CsA and Dydrogesterone.

SECONDARY OUTCOMES:
The difference in the rate of miscarriage between patients with recurrent miscarriage treated with CsA and Dydrogesterone. | Up to 36 months
  The difference in the rates of miscarriage (pregnancy loss before 20 weeks gestation) between patients assigned oral CsA and Dydrogesterone.
Fetal death | Up to 36 months
  The difference in the rates of fetal death (fetal death after 20 weeks of gestational age) between patients assigned oral CsA and Dydrogesterone.
The difference in the rate of premature delivery between patients treated with CsA and Dydrogesterone. | Up to 36 months
  The difference in the rates of premature delivery (deliveries with gestational age less than 37 weeks) between patients assigned oral CsA and Dydrogesterone.
Congenital malformations | Up to 36 months
  The difference in the rates of congenital malformations between patients assigned oral CsA and Dydrogesterone.
Maternal outcomes: morbidity of infectious disease | Up to 36 months
  The difference of morbidity of infectious disease in pregnancy between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dajin Li, MD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YH, Ma YL, Ma L, Mao JL, Zhang Y, Du MR, Li DJ. Cyclosporine A improves adhesion and invasion of mouse preimplantation embryos via upregulating integrin beta3 and matrix metalloproteinase-9. Int J Clin Exp Pathol. 2014 Mar 15;7(4):1379-88. eCollection 2014. PMID 24817934
- [Background] Wang SC, Yu M, Li YH, Piao HL, Tang CL, Sun C, Zhu R, Li MQ, Jin LP, Li DJ, Du MR. Cyclosporin A promotes proliferating cell nuclear antigen expression and migration of human cytotrophoblast cells via the mitgen-activated protein kinase-3/1-mediated nuclear factor-kappaB signaling pathways. Int J Clin Exp Pathol. 2013 Sep 15;6(10):1999-2010. eCollection 2013. PMID 24133577
- [Background] Piao HL, Wang SC, Tao Y, Zhu R, Sun C, Fu Q, Du MR, Li DJ. Cyclosporine A enhances Th2 bias at the maternal-fetal interface in early human pregnancy with aid of the interaction between maternal and fetal cells. PLoS One. 2012;7(9):e45275. doi: 10.1371/journal.pone.0045275. Epub 2012 Sep 27. PMID 23028901
- [Background] Wang SC, Tang ChL, Piao HL, Zhu R, Sun Ch, Tao Y, Fu Q, Li DJ, Du MR. Cyclosporine A promotes in vitro migration of human first-trimester trophoblasts via MAPK/ERK1/2-mediated NF-kappaB and Ca2+/calcineurin/NFAT signaling. Placenta. 2013 Apr;34(4):374-80. doi: 10.1016/j.placenta.2013.01.009. Epub 2013 Feb 11. PMID 23410723
- [Background] Zhao HB, Tang CL, Hou YL, Xue LR, Li MQ, Du MR, Li DJ. CXCL12/CXCR4 axis triggers the activation of EGF receptor and ERK signaling pathway in CsA-induced proliferation of human trophoblast cells. PLoS One. 2012;7(7):e38375. doi: 10.1371/journal.pone.0038375. Epub 2012 Jul 27. PMID 22848341
- [Background] Tang CL, Zhao HB, Li MQ, Du MR, Meng YH, Li DJ. Focal adhesion kinase signaling is necessary for the Cyclosporin A-enhanced migration and invasion of human trophoblast cells. Placenta. 2012 Sep;33(9):704-11. doi: 10.1016/j.placenta.2012.06.007. Epub 2012 Jul 4. PMID 22766276
- [Background] Du MR, Zhou WH, Piao HL, Li MQ, Tang CL, Li DJ. Cyclosporin A promotes crosstalk between human cytotrophoblast and decidual stromal cell through up-regulating CXCL12/CXCR4 interaction. Hum Reprod. 2012 Jul;27(7):1955-65. doi: 10.1093/humrep/des111. Epub 2012 Apr 11. PMID 22495096
- [Background] Du MR, Zhou WH, Dong L, Zhu XY, He YY, Yang JY, Li DJ. Cyclosporin A promotes growth and invasiveness in vitro of human first-trimester trophoblast cells via MAPK3/MAPK1-mediated AP1 and Ca2+/calcineurin/NFAT signaling pathways. Biol Reprod. 2008 Jun;78(6):1102-10. doi: 10.1095/biolreprod.107.063503. Epub 2008 Mar 5. PMID 18322274
- [Background] Zhou WH, Dong L, Du MR, Zhu XY, Li DJ. Cyclosporin A improves murine pregnancy outcome in abortion-prone matings: involvement of CD80/86 and CD28/CTLA-4. Reproduction. 2008 Mar;135(3):385-95. doi: 10.1530/REP-07-0063. PMID 18299432
- [Background] Du MR, Zhou WH, Yan FT, Zhu XY, He YY, Yang JY, Li DJ. Cyclosporine A induces titin expression via MAPK/ERK signalling and improves proliferative and invasive potential of human trophoblast cells. Hum Reprod. 2007 Sep;22(9):2528-37. doi: 10.1093/humrep/dem222. Epub 2007 Jul 18. PMID 17636278
- [Background] Zhou WH, Du MR, Dong L, Zhu XY, Yang JY, He YY, Li DJ. Cyclosporin A increases expression of matrix metalloproteinase 9 and 2 and invasiveness in vitro of the first-trimester human trophoblast cells via the mitogen-activated protein kinase pathway. Hum Reprod. 2007 Oct;22(10):2743-50. doi: 10.1093/humrep/dem097. Epub 2007 Jun 12. PMID 17566014
- [Background] Du MR, Dong L, Zhou WH, Yan FT, Li DJ. Cyclosporin a improves pregnancy outcome by promoting functions of trophoblasts and inducing maternal tolerance to the allogeneic fetus in abortion-prone matings in the mouse. Biol Reprod. 2007 May;76(5):906-14. doi: 10.1095/biolreprod.106.056648. Epub 2007 Jan 17. PMID 17229932